CLINICAL TRIAL: NCT03290040
Title: Identification of Predictors for Early Cognitive Decline: a Longitudinal Cohort Study in Men Born in 1953
Brief Title: Identification of Predictors for Early Cognitive Decline in Men
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Martin Lauritzen, Professor, Consulting, Rigshospitalet, Denmark
Other Study IDs: H-1-2014-032
Record Dates: First submitted 2015-11-18; First posted 2017-09-21 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Healthy Test Persons; Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples with DNA

GROUPS / COHORTS (2):
- Metropolit Cohort: Danish birth cohort of men born in 1953 in the Metropolitan area of Copenhagen. These test-persons are divided into two groups based on performance in cognitive tests at late midlife compared to young adulthood; Positive expected performance and negative expected performance and sampled from a birth cohort of 11.532 men.
- Herlev Hospital, Memory Clinic: Persons from the Memory Clinic at Herlev Hospital. These subjects are diagnosed with either MCI or AD.

SUMMARY:
The research program explores how aging influences brain function in test-persons from a Danish birth cohort of men born in 1953.

DETAILED DESCRIPTION:
The research program explores how ageing influences brain function in healthy test-persons from a Danish birth cohort of men born in 1953 in the Metropolitan area of Copenhagen. These test-persons are divided into two groups based on performance in cognitive tests at late midlife compared to young adulthood; Positive expected performance and negative expected performance and sampled from a birth cohort of 11.532 men.

Additionally, persons diagnosed with either MCI or AD will be included from the Memory Clinic at Herlev Hospital.

Researchers aim to identify factors earlier in life that affects or predict changes in cognitive function, specifically of cognitive decline in order to predict healthy vs unhealthy cognitive ageing, including progression to possible dementia. The objective is to be able to predict cognitive decline in ageing.

During the years of data collection, approximately 550 participants will be included and examined.

The examinations include:

* Cognitive test including Cambridge Neuropsychological test automated Battery (CANTAB);
* Sleep
* Life events
* Depression questionnaire
* Blood sample analysis including functional analyses of mitochondria and gene analyses such as genome scanning, SNP analysis
* ApoE ε-type
* Structural and functional changes in the brain measured with magnetic resonance (fMRI)
* Electroencephalography (EEG) recordings of electrical activity and visual attention
* PET-scan (Amyloid and FDG)

The results from these studies will hopefully point to new avenues for intervention in order to change the course of brain ageing

ELIGIBILITY:
Inclusion Criteria:

* Participants who have participated in the Metropolit study and the Copenhagen Aging and Midlife Biobank project
* Participants who have been informed about the project and who have signed the informed consent form

Exclusion Criteria:

* Persons who have been asked to participate in the past and have rejected
* Reduced ability to understand project information
* Reduced ability to complete the examinations
* Abuse of alcohol, psychedelic drugs or habit-forming drugs
* Certain neurological disorders
* Certain neurological, mental or psychiatric diagnoses
* Certain depressive diseases
* Former traumatic brain injury
* Contraindication for MR scanning
* Pathological MR result
* Persons that do not like to be informed about a possible pathological result

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish birth cohort of 11.532 men born in 1953 in the Metropolitan area of Copenhagen.
  Only men who have participated in the Copenhagen Aging and Midlife Biobank project are considered.
  Persons from the Memory Clinic at Herlev Hospital will be included in the period 2020-2021. These individuals are diagnosed with either MCI or AD.
Sampling Method: Non-Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Gamma band EEG power during evoked potentials correlates to cognitive decline | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Visual and auditory evoked potentials are elicited in the brain using flickering visual stimuli and amplitude-modulated tones, respectively. The potentials are recorded through scalp electroencephalography (EEG), using a 64-channel EEG cap. A measure of cognitive decline is approximated using intelligence test scores collected at three distinct times in the lifespan of the subject, as well as other clinical cognitive tests sensitive to aging effects
Alpha band EEG-power during evoked potentials correlates to cognitive decline | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Visual evoked potentials are elicited in the brain using flickering visual stimulus. The potentials are recorded through scalp electroencephalography (EEG), using a 64-channel EEG cap. A measure of cognitive decline is approximated using intelligence test scores collected at three distinct times in the lifespan of the subject, as well as other clinical cognitive tests sensitive to aging effects
Examination of how visual attention effects cognitive deterioration. | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  The accuracy of reporting shown isoluminant letters of the patient is compared to speed of processing (ms), IQ and short term memory function.
Clarification of how processing speed (ms), short term memory and visual perceptive threshold effect cognitive capacity. | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Relating brain states to attentional functions by linking visual event-related potentials measured with EEG to specific attentional functions derived from behavioural testing
Changes in mitochondrial respiration as predictor of cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Microstructural parameters, derived from diffusion tensor imaging as predictor of cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Correlation between basal ganglia volumes and structure and cognitive functions | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive composite scores are based on CANTAB as well as paper and pencil tests. Basal ganglia volumes are based on automatic segmentation procedures. Basal ganglia microstructure and iron content will be estimated using quantitative susceptibility imaging
Correlation between patterns of brain perfusion and patterns of cognitive function | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive composite scores are based on CANTAB as well as paper and pencil tests. Brain perfusion will be measured with arterial spin labeling, and the analysis performed using multivariate techniques
Correlation between Subjective sleep quality and patterns of cognitive function | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive functions are based on CANTAB as well as paper and pencil tests. Sleep quality is measured using the self-report questionnaire Pittsburgh Sleep quality Index (PSQI).
Objective sleep measures: Sleep stages as determined by standard international scoring and quantitated measures using - spectral analysis from sleep EEG in relation to cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Effects of demographic, social and health predictors on change in cognitive function from young adulthood to late midlife | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive composite score (based on CANTAB, paper- and pencil tests)
Correlation between daytime sleepiness and patterns of cognitive function | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive functions are based on CANTAB as well as paper and pencil tests. Daytime sleepiness is measured using the Epworh Sleepiness Scale (ESS) questionnaire.
FDG - PET | This examination will be performed in 2020-2021.
  FDG - PET scan uses a special radioactive glucose-analogue tracer which the body uptake similarly to normal glucose. This allows us to investigate how well an individual can uptake glucose in relevant brain areas and thereby how well they increase the metabolism and activity in these brain areas when stimulated.
  With this method, we can see how the brain is working and detect any abnormalities.
PIB - PET | This examination will be performed in 2020-2021.
  PIB - PET scan uses special radioactive tracers that highlight amyloid protein plaques in the brain, which are a hallmark of Alzheimer's disease. This scanning will allow us to see the distribution of Amyloid plaques in the cohort and to test for correlation with cognitive decline.

SECONDARY OUTCOMES:
Gamma band EEG power distribution across the scalp during simultaneous auditory and visual stimulation correlates to cognitive decline | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Visual and auditory evoked potentials are elicited in the brain using a paradigm that presents a visual stimulus and an auditory stimulus simultaneously. The potentials are recorded through scalp electroencephalography (EEG), using a 64-channel EEG cap. A measure of cognitive decline is approximated using intelligence test scores collected at three distinct times in the lifespan of the subject
Change of source location of gamma band EEG power of visual evoked potentials correlates to cognitive decline | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Visual evoked potentials are elicited in the brain using flickering visual stimulus. The potentials are recorded through scalp electroencephalography (EEG), using a 64-channel EEG cap. A measure of cognitive decline is approximated using intelligence test scores collected at three distinct times in the lifespan of the subject, as well as other clinical cognitive tests sensitive to aging effects
The investigators would like to describe how visual attention correlates with the background EEG recorded before the examination. | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Linking functional effects of prestimulus alpha power measured by EEG to perception accuracy
Change in levels of reactive oxygen species in PBMCs quantified by flow cytometry after application of dedicated fluorophores as predictor of cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Change in levels of mitochondrial bioenergetics in PBMCs using the Seahorse XF24 extracellular flux analyser as predictor of cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Change of levels of whole cell dNTP levels in PBMCs using polymerase extension assay and by quantification of tritiated nucleotides by scintillation counting as predictor of cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Change of mutation frequency of mitochondrial DNA using deep sequencing as predictor of cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Change of mtDNA copy number by qPCR as predictor of cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Correlation between regional cortical thickness and cognitive parameters | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive composite scores are based on CANTAB as well as paper and pencil tests. Cortical thickness will be analysed using FreeSurfer or similar software, and the analysis performed using multivariate techniques
Correlation between regional cortical surface and cognitive parameters | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive composite scores are based on CANTAB as well as paper and pencil tests. Cortical surface will be analysed using FreeSurfer or similar software, and the analysis performed using multivariate techniques
Correlation between macrostructural parameters and candidate genes | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Macrostructural parameters will be derived from segmentation of T1-weighted images. The statistical analysis will consider macrostructural parameters as a possible mediator of common genetic variants upon cognition. Candidate genes will be selected due to their relation to 1) cardiovascular function and disease 2) oxidative stress, longevity and ageing and 3) memory and intelligence.
Correlation between microstructural parameters and candidate genes | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Microstructural parameters will be derived from diffusion tensor imaging. The statistical analysis will consider microstructural parameters as a possible mediator of common genetic variants upon cognition. Candidate genes will be selected due to their relation to 1) cardiovascular function and disease 2) oxidative stress, longevity and ageing and 3) memory and intelligence.
Correlation between macrostructural parameters and cognition | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Macrostructural parameters will be derived from segmentation of T1-weighted images. Cognitive composite scores are based on CANTAB as well as paper and pencil test.
Correlation between microstructural parameters and cognition | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Microstructural parameters will be derived from diffusion tensor imaging. Cognitive composite scores are based on CANTAB as well as paper and pencil test.
Correlation between cognition and candidate genes | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive composite scores are based on CANTAB as well as paper and pencil test.Candidate genes will be selected due to their relation to 1) cardiovascular function and disease 2) oxidative stress, longevity and ageing and 3) memory and intelligence.
Correlation between sleep stages and microstructural parameters. | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Sleep stages will be determined by standard international scoring and quantitated measures using spectral analysis from sleep EEG. Microstructures will be measured with MRI.
Correlation between sleep stages and regional volumes. | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Sleep stages will be determined by standard international scoring and quantitated measures using spectral analysis from sleep EEG. Regional volumes will be measured with MRI.
Autonomic activity as measured by electrocardiography determined from the polysomnography during wakefulness and sleep in relation to cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Presence of REM Sleep muscle activity (REM sleep without atonia (RSWA), REM Behavior disorder(RBD)) in relation to cognitive impairment | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
Cognitive correlates of cognitive change | Participant is recruited and measured once at the examination day and reexamined every 5 year as long as the project is running and includes the measurement, expected up to 10 years
  Cognitive composite score (based on CANTAB, paper- and pencil tests)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J Lauritzen, Prof, Principal Investigator — Dept. of Clinical Neurophysiology, Rigshospitalet - Glostrup; Martin J Lauritzen, Prof, Principal Investigator — Dept. of Clinical Neurophysiology, Rigshospitalet - Glostrup, Neuronal Signalling Lab, Center for Neuroscience, and Center for Healthy aging, University of Copenhagen
Locations (1):
- Dept. of Clinical Neurophysiology, Department of Clinical Biochemistry and Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet - Glostrup, Glostrup Municipality, Denmark